CLINICAL TRIAL: NCT06298422
Title: Addressing Race-Based Limitations in Pulse Oximetry Through Colorimeter or Spectrophotometer-Integrated Corrections
Brief Title: Oxygen Saturations Across Tones of Skin
Acronym: O2SATS
Status: Enrolling by invitation | Type: Observational
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Shannon Cotton, Principal Investigator, University of California, San Diego
Other Study IDs: 806433
Record Dates: First submitted 2024-02-22; First posted 2024-03-07 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Generalised Melanin Pigmentation; Pulse Oximetry

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Pulse oximetry, or SpO2, is a vital sign used across healthcare systems to gauge how much oxygen blood is carrying as a percentage of the maximum it could carry. Recent research has suggested that current SpO2 monitors may inaccurately report high SpO2 in patients with darker skin tones when the actual oxygenation is at unsafe, low levels. Additionally, this new research suggests as the SpO2 levels decrease, the risk of occult hypoxia rises. The investigators hypothesize melanin interferes with the pulse oximetry accuracy. Investigators will use spectrophotometry to measure melanin indices and other variables to test this hypothesis.

ELIGIBILITY:
Inclusion criteria:

1. >18 years old
2. Any gender
3. Any ethnic background
4. Admitted to UC San Diego La Jolla or Hillcrest campus ICU
5. Mechanically ventilated
6. Has a clinical ABG ordered by the critical care team responsible for clinical care

Exclusion Criteria a. <18 years old b. Medical history of or acute diagnosis of sickle cell disease c. Normally protected individuals under 45 CFR 46 (pregnant individuals, prisoners, and children)

-

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critically ill patients on mechanical ventilation.
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Difference observed between SpO2 and SaO2. | Through study completion, approximately one year
  Arterial Blood Gas
Melanin Index | Through study completion, approximately one year
  Spectrophotometry

CONTACTS AND LOCATIONS:
Locations (1):
- UCSD Health, San Diego, California, United States